CLINICAL TRIAL: NCT00020800
Title: Phase II Study of Combination Rituxan (Rituximab, Mabthera) and Fludarabine Therapy in Lymphoplasmacytic Lymphoma (Waldenstrom's Macroglobulinemia)
Brief Title: Rituximab Plus Fludarabine in Treating Patients With Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068714; UCLA-0101063; NCI-G01-1960
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Rituximab; fludarabine phosphate

INTERVENTIONS:
Biological: rituximab
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different way to stop cancer cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab plus fludarabine in treating patients who have Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response and time to treatment failure in patients with Waldenstrom's macroglobulinemia treated with rituximab and fludarabine.
* Determine the toxicity of this regimen in these patients.
* Determine if molecular remissions are achievable in patients attaining a clinical complete response when treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV over 3-6 hours once weekly on weeks 1-4, 17, 18, 30, and 31 and fludarabine IV over 10-30 minutes once daily for 5 days on weeks 5, 9, 13, 19, 23, and 27.

Patients are followed at least every 2 months for 2 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Waldenstrom's macroglobulinemia
* CD20 positive by bone marrow immunohistochemistry or flow cytometry
* Presence of monoclonal paraprotein
* IgM level at least 2 times upper limit of normal (ULN)

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* At least 6 months

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 25,000/mm^3

Hepatic:

* Bilirubin less than 2.5 times ULN
* SGOT less than 2.5 times ULN

Renal:

* Creatinine less than 2.5 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after study
* No serious comorbid disease
* No uncontrolled bacterial, fungal, or viral infection
* No other active malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior rituximab
* No prior nucleoside analogue therapy

Chemotherapy:

* At least 30 days since prior chemotherapy

Endocrine therapy:

* At least 30 days since prior steroid therapy
* No concurrent corticosteroids

Radiotherapy:

* At least 30 days since prior radiotherapy

Surgery:

* Not specified

Other:

* No more than 2 prior courses of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2001-09; Primary Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (18):
- United States (14):
  - Arizona Cancer Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Tuft-New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
- Huddinge University Hospital, Stockholm, Sweden
- Saint Bartholomew's Hospital, London, England, United Kingdom

REFERENCES:
- [Result] Treon SP, Branagan AR, Ioakimidis L, Soumerai JD, Patterson CJ, Turnbull B, Wasi P, Emmanouilides C, Frankel SR, Lister A, Morel P, Matous J, Gregory SA, Kimby E. Long-term outcomes to fludarabine and rituximab in Waldenstrom macroglobulinemia. Blood. 2009 Apr 16;113(16):3673-8. doi: 10.1182/blood-2008-09-177329. Epub 2008 Nov 17. PMID 19015393